CLINICAL TRIAL: NCT02195076
Title: A Clinical Study Design to Evaluate the Specificity and Sensitivity of Our Novel System for Detection of Breast and Lung Cancer by Odor Signature
Brief Title: Non Invasive Detection of Lung and Breast Cancer by Odor Signature
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BioSense Medical LTD (Industry)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0695-13-SMC
Record Dates: First submitted 2014-07-16; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Lung Cancer; Breast Cancer
Keywords: Lung cancer; Breast Cancer; Biosensors; Volatile Organic Compounds; Odor; Urine Sample; Exhaled Breath Samples
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — urine samples and exhaled breath samples

GROUPS / COHORTS (3):
- Breast Cancer patients
  Interventions: Other: non-invasive detection of cancer odor
- Lung cancer patients
  Interventions: Other: non-invasive detection of cancer odor
- Healthy controls
  Interventions: Other: non-invasive detection of cancer odor

INTERVENTIONS:
Other: non-invasive detection of cancer odor — The odor VOCs of the specimens will be subjected to our system for detection by the biosensors. If the sample is cancerous the biosensors will report it (YES signal). If the sample s not cancerous, the biosensors will not report it (NO signal).

SUMMARY:
The investigators have developed an early detection solution for lung and breast cancer. A system which can distinguish between different medical odors based on biosensors. Our product is user-friendly noninvasive, nonradioactive and nontoxic to the patients. The technology enables a high level of sensitivity and provides users with a quick lab response and a simple yes or no answer.

The aim of this study is to contribute and detect the patient at the earliest possible stage, in a noninvasive, nonradioactive and nontoxic way. Exhaled breath and urine samples are a promising approach towards future possible lung and breast cancer screening method.

DETAILED DESCRIPTION:
Early detection of cancer can dramatically improve the survival chances. to date, there is no efficient diagnostic tool for detection of lung cancer in early stages. Regarding breast cancer, the common screening tool us mammography, which suffer from low sensitivity and high false positive. Thus, there is an urgent need for developing a screening tool for early stages lung and breast cancer.

The sense of smell depends on the ability of specialized sensory cells of the nose to perceive volatile compounds (VOCs). Diseases such as infections and malignancies can be associated with changes in host metabolism, accompanied by production of different VOCs, and thus a different odor. Several studies have shown that different cancers secrete different VOCs, thus produce different smell.

We have developed a system which uses biosensors that can scent the VOCs that lung and breast cancer cell produce, thus distinguish between healthy control and lung or breast cancer. These biosensors can detect low stages lung and breast cancer.

Patients will supply urine samples and exhaled breath samples using a kit that we will supply. The samples will be shipped to our lab, where they will be processed and the VOCs will be separated from the head space of the samples. The biosensors will be exposed to the VOCs samples and will report whether the specific sample id cancerous (lung or breast) or not.

The Data will be collected from all samples and statistical analysis will be calculated, in order to test the specificity and sensitivity of our biosensors to detect cancerous samples.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Lung Cancer patients
* Diagnosed Breast Cancer patients

Exclusion Criteria:

* Cancer patients who were treated using chemotherapy
* Cancer patients who were treated using radiation
* Cancer patients who were treated using biological treatments
* Cancer patients who were treated with chemotherapy
* Cancer patients who were treated with any anti- cancer therapies
* Cancer patients who use drugs that affect the immune system

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast Cancer patient after diagnosis. Lung Cancer patients after diagnosis. Healthy controls, matching gender and age.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of our biosensors in lung and breast cancer detection | 3 years
  We will measure the ability of our biosensors to detect lung and breast cancer in urine samples from patients. Each urine sample will be subjected to 5 biosensors. If 3 out of 5 will report positively, the sample will be marked as cancerous. Each type of cancer (lung or breast) will be detected by different groups of biosensors, trained specifically to detect the specific cancer type.
  After the data of the detections will be collected, statistical analysis will be calculated in order to evaluate the sensitivity and specificity of our biosensor in cancer detection.

SECONDARY OUTCOMES:
Testing the ability of our biosensors to distinguish between different sub- types of breast and lung cancer. | 3 years
  After the collection of the detection data (primary outcome measure), we will compare it to the patients data records (in terms of staging, CT, pathology, biological markers etc.) and evaluate whether our biosensors can detect different sub- types of lung and breast cancer in different sensitivity and specifity.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Hashomer, Ramat- Gan, Israel